# STATISTICAL ANALYSIS PLAN

#### LA48-0215

A Dose-Ranging Study of the Efficacy, Safety, and Pharmacokinetics of Deferiprone Delayed Release Tablets in Patients with Parkinson's Disease

Final Version 1.0

Prepared by

Feng Zhao

Scientific Leader, Biostatistics

ApoPharma Inc.

18 JUN 2019

Date (DD-MMM-YYYY)

### CONFIDENTIAL DOCUMENT

The information contained in this Statistical Analysis Plan is confidential and is the property of ApoPharma Inc. Do not release information from this Statistical Analysis Plan without written permission of ApoPharma Inc.

### Approvals

Caroline Fradette, PhD Director, Clinical Research ApoPharma Inc., Canada

Anna Rozova, MD Director, Medical Safety ApoPharma Inc., Canada

Yu-Chung Tsang, PhD Chief Scientific Officer Biopharmaceutics and Biostatistics Apotex Inc., Canada

Date (DD-MMM-YYYY)

Date (DD-MMM-YYYY)

## **Table of Contents**

| | Title | e page | | 1 |
|---|---|---|---|---|
| | | | ntents | |
| | | | reviations | |
| 1 2 | | | ntives | |
| <u></u> | 2.1 | • | ry Objective | |
| | 2.2 | | dary Objectives | |
| | 2.3 | | ratory Objectives | |
| 3 | | | | |
| | 3.1 | | Design and Randomization | |
| | 3.2<br>3.3 | <ul><li>3.2 Determination of Sample Size and Study Power</li><li>3.3 Analysis Populations</li></ul> | | |
| | 3.4 | • | m Analysis | |
| | 3.5 | | ng Data Handling and Derivation Rules | |
| | 3.6 | | ical Software and Level of Significance | |
| 4 | | | analyses | |
| | 4.1 | | t Disposition and Drug Exposure | |
| | 4.2 | | t Characteristics | |
| | | 4.2.1 | Demographics | |
| | | 4.2.2 | Medical History | 12 |
| | | 4.2.3 | Prior Medications | 12 |
| | 4.3 | Effica | cy Analyses | 12 |
| | | 4.3.1 | Primary Efficacy Endpoint | 12 |
| | | 4.3.2 | Secondary Efficacy Endpoints | 13 |
| | | 4.3.3 | Exploratory Efficacy Endpoints | 14 |
| | | 4.3.4 | Exploratory Analyses/Sensitivity Analysis | 15 |
| | 4.4 | Safety | Analyses | 15 |
| | | 4.4.1 | Adverse Events | 16 |
| | | 4.4.2 | Vital Signs and Weight | 18 |
| | | 4.4.3 | 12-Lead ECG | 18 |
| | | 4.4.4 | Biochemistry, Hematology and Urinalysis | 18 |
| | | 4.4.5 | Concomitant Medications | 18 |
| | | 4.4.6 | Suicidality | 19 |
| | | 4.4.7 | Treatment Compliance | 19 |

| 5 | Listing of Tables and Figures20 |
|---|---------------------------------|
| | Data Listings25 |
| | Table Shells 27 |

#### List of Abbreviations

ADR Adverse Drug Reaction

AE Adverse Event

ANOVA Analysis of Variance

AUCss Area under the concentration-time curve at steady state

CI Confidence Interval
Cmax Maximum Concentration
COMT Catechol O-methyltransferase

C-SSRS Columbia Suicide Severity Rating Scale
DDFM Denominator Degrees of Freedom Method

DFP Deferiprone
DR Delayed Release
ECG Electrocardiogram

eCRF electronic Case Report Form

ITT Intent-to-treat

KR Kenward and Roger's method LOCF Last Observation Carried Forward

LSM Least Square Mean

MDS-UPDRS Movement Disorder Society-Unified Parkinson's Disease Rating

Scale

MedDRA Medical Dictionary for Regulatory Activities

mg Milligram

MMRM Mixed-Effect Model Repeated Measure

MOA Mechanism of Action

MoCA Montreal Cognitive Assessment

PD Pharmacodynamics
PK Pharmacokinetics
PP Per protocol
PT Preferred Term

SAE Serious Adverse Event SD Standard Deviation SOC System Organ Class

#### 1 Introduction

This document outlines the statistical analysis plan for the efficacy and safety analysis for the clinical trial LA48-0215 sponsored by ApoPharma Inc.

#### 2 Study Objectives

#### 2.1 Primary Objective

• To evaluate the efficacy of four different dosages of deferiprone delayed release (deferiprone-DR) tablets in patients with Parkinson's disease

#### 2.2 Secondary Objectives

- To evaluate the safety and tolerability of deferiprone-DR tablets in patients with Parkinson's disease
- To evaluate the pharmacokinetics of deferiprone-DR tablets in a subset of study participants
- To evaluate the relationship between the pharmacokinetics and pharmacodynamics of deferiprone-DR tablets

#### 2.3 Exploratory Objectives

- To determine whether the efficacy responses to deferiprone differ depending on the genotype of certain enzymes that are implicated in Parkinson's disease
- To determine whether the efficacy responses to deferiprone are correlated with ceruloplasmin levels or ceruloplasmin ferroxidase activities

#### 3 Methods

#### 3.1 Study Design and Randomization

This is a multi-center, randomized, double-blind, placebo-controlled, dose-ranging study in 140 patients who had been diagnosed with typical Parkinson's disease within the last 3 years and were taking antiparkinsonian medication at enrollment. Screening was conducted within 30 days prior to the start of dosing. At baseline, eligible participants were randomized to one of four dosage cohorts, and within each cohort were further

randomized in a 4:1 ratio to receive either active product (n=28) or placebo (n=7). Thus, a total of 112 patients received one of the four dosages of deferiprone, and a total of 28 received placebo. The assigned study product was taken twice-daily (b.i.d.), at least 8 hours apart, for 9 months. Dosages were as follows:

- Cohort 1: 300 mg deferiprone delayed release tablets (n=28) or placebo (n=7)
- Cohort 2: 600 mg deferiprone delayed release tablets (n=28) or placebo (n=7)
- Cohort 3: 900 mg deferiprone delayed release tablets (n=28) or placebo (n=7)
- Cohort 4: 1200 mg deferiprone delayed release tablets (n=28) or placebo (n=7)

Patients returned to the site at Months 1, 2, 3, 4, 5, 6, and 9, and received a follow-up telephone call at Month 10. Safety was assessed at each site visit and at the follow-up call; efficacy measures were assessed at baseline and Months 3, 6, and 9; and sparse pharmacokinetics (PK) sampling was done on all patients at baseline and Month 3. In addition, an optional subset of 16 patients underwent extensive blood sampling for PK analysis at Month 1, and an optional subset of 18 patients each provided one sample of cerebrospinal fluid (CSF) for drug level analysis at Month 3. (No selection was done to enroll these subsets: all patients were asked if they were willing to provide either or both of these types of samples, and they were enrolled as they came until the total number of subjects was reached for each subset.) For safety reasons, all patients had their absolute neutrophil count monitored weekly after the start of dosing, at either the study site or a local laboratory. Any patient whose regimen of antiparkinsonian medication was changed, including a change in dosage, would be withdrawn from the trial.

Any patient who withdrew before completing treatment was requested to return within one month for an Early Termination visit, at which time the procedures normally scheduled for the Month 9 visit were conducted.

#### 3.2 Determination of Sample Size and Study Power

There was no formal sample size and power calculation for this Phase II dose-finding study.

#### 3.3 Analysis Populations

Four study populations for analysis are defined: Intent-to-Treat (ITT), Per-Protocol (PP), Safety, and Pharmacokinetics/Pharmacodynamics (PK/PD). For efficacy, all endpoints will be analyzed for the ITT population, which represents the primary analysis population, and the primary efficacy endpoint will additionally be analyzed for the PP population, which represents the secondary analysis population.

#### **ITT Population**

The ITT population is defined as all randomized patients who received at least one dose of study drug and havea baseline and at least one post-baseline efficacy assessment for the primary endpoint. All efficacy endpoints will be analyzed for the ITT population.

### PP Population

The PP population is defined as all randomized patients who completed the study, have no major protocol violations, and have an efficacy assessment for the primary endpoint at the end of the study. Prior to database lock, protocol violations will be reviewed for their seriousness, and patients with major violations will be excluded from the PP population. The only endpoint that will be analyzed for the PP population is the the primary efficacy endpoint.

### **Safety Population**

The Safety population will include all randomized patients who received at least one dose of study drug.

### PK/PD Population

The Pharmacokinetics/Pharmacodynamics (PK/PD) population will include all patients who provided sufficient PK data to derive at least one PK parameter. Detailed analyses on PK assessments will be included in separate statistical analysis plan.

#### 3.4 Interim Analysis

No interim analysis is planned or conducted.

#### 3.5 Missing Data Handling and Derivation Rules

For safety data and PD data, all analyses will be based on observed cases (OC). No imputation will be performed on missing data.

For all efficacy measures but one (time elapsed until rescue medication), when there are missing total scores, missing data will be assumed to be missing at random (MAR). A Mixed-Effect Model Repeated Measure (MMRM) model will be used as the primary analysis method, and the analyses will be based on observed cases. A sensitivity analysis will be conducted for the primary efficacy endpoint, with missing data being imputed as follows. In cases where early termination was due to either worsening of disease conditions or inadequate efficacy of the drug (as documented in the case report form), the "worst score" method will be used to fill in missing data. With this method, for the placebo group, the average change score of the placebo group at a particular visit will be used to impute any missing data at that visit, while for the active group, the worst change score of all patients at that visit will be used. In cases where early termination was due to some other reason, such as a missed visit, the last observation carried forward (LOCF)

method will be used to fill in the missing data. For Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score, a score will be obtained for each part and a total score will be calculated by adding the score of each part. For each part, one would simply add the score obtained for all questions. If there is a missing answer, the score for this part will be handled as below:

- $\circ$  (A x B) / C = D
- o Where:
  - A = sum of all item score recorded in a specific part
  - B = number of total items in a specific part
  - C = number of item with actual score in specific part
  - D = final calculated valid Part score

For example, if a part has 13 items and only 12 items have been rated, one will get the sum of these 12 items, multiply it by 13 and dividing this by 12.

However, for an imputed score to be valid for a specific part, the below maximum of item missed per part cannot be exceeded:

- Part I: max of 2 missing items
- Part II: max of 3 missing items
- Part III: max of 9 missing items
- Part IV: max of 1 missing items

If there are more than the maximum number of item missed in a part, the total score for that part will not be imputed and will be left as missing.

For Montreal Cognitive Assessment (MoCA) test score, the missing component score will be assigned a score of zero by the rater so it is expected the number of missing component score will be minimal. If there is a missing component score, it will be imputed by the LOCF method before the total score is calculated.

Date of exposure will be defined as Day 1 for all duration calculations. For example, age at entry will be calculated as the integer value of the expression:

Floor(date of exposure – date of birth) / 365.25

Time in months will be derived by dividing the time in days by 30.4.

#### 3.6 Statistical Software and Level of Significance

All statistical analyses will be performed using SAS (version 9.3 or higher) on the Windows operating system. The null hypotheses tested are that there is no difference in true parameter between comparison groups, unless otherwise stated. A two-sided p-value of 0.05 will be used as the significance level for the determination of statistical significance in all statistical tests.

#### 4 Statistical Analyses

Data from all patients who were randomized to receive placebo will be combined into one group for the efficacy and safety analyses. Thus, there will be a total of 5 treatment groups: the placebo group and the 300 mg, 600 mg, 900 mg, and 1200 mg deferiprone groups. Descriptive statistics will be used to summarize continuous variables, while frequency and percentage will be presented for each discrete variable. Where applicable, analysis of variance (ANOVA) will be used to compare means, and Fisher's exact test will be used to compare proportions.

As patients may not attend each study visit within the specified time window, efficacy data will be classified into scheduled visits according to the time elapsed from the first dose of medication (date of exposure) to the date of assessment, as follows:

Month 3 visit: 0 to < 4.5 months

Month 6 visit: 4.5 to < 7.5 months

Month 9 visit: 7.5 to < 10.5 months

The calculation of time elapsed from the date of exposure to the date of assessment is done as follows:

Time elapsed = (date of sample assessment) – (date of exposure) +1

The resulting time elapsed will be expressed in months. If this results in overlap in visits, the average value of the same visits will be used in the analysis.

For all continuous efficacy outcomes except for time elapsed until rescue medication (addressed below), a Mixed-Effect Model Repeated Measure (MMRM) model will be used as the primary analysis method to assess the effect of deferiprone on change from baseline to Month 9. The MMRM model will include the baseline value of the outcome as a covariate and treatment group and visit as the main factors. Baseline value is the value collected the closest prior to baseline visit.

The MIXED procedure in SAS will be used for the MMRM model analysis. Data from each patient at different visits will be considered repeated measures. A first-order

autoregressive (AR) covariance structure will be used to model the correlation between repeated measures within the same patient, and Kenward and Roger's method will be used to estimate the denominator degrees of freedom (DDFM). The Least Square Mean (LSM) and 95% confidence interval (CI) of the LSM difference will be calculated by the LSMEANS statement.

A sample SAS code for the MMRM model is shown in the box below:

```
proc mixed;
  class TREAT USUBJID VISIT;
  model CHG=TREAT VISIT TREAT*VISIT BASE/solution ddfm=kr;
  repeated VISIT/ subject=USUBJID type=ar(1);
  lsmeans TREAT*VISIT / diff cl;
run;
```

where TREAT is the discrete variable for treatment group, USUBJID represents the patient ID, VISIT is the discrete variable representing the scheduled study visit after the baseline visit, CHG is the change in value of efficacy outcome from baseline to the scheduled visit, and BASE is the baseline value of efficacy outcome.

If the treatment effect is found to be statistically significant, each deferiprone group will be compared to the placebo group to assess the treatment effect at each deferiprone dose level using the SAS code for MMRM model as presented above. Linear regression analysis will be employed to assess the dose-response relationship through a linear regression model, with the change at the study end as the dependent variable and the treatment dose as the continuous variable. If a statistically significant relationship exists between deferiprone dose and an efficacy outcome, the dose-response relationship will be further assessed and reported through pairwise comparison of each dose level to the next lower dose level: 1200 mg vs. 900 mg, 900 mg vs. 600 mg, and 600 mg vs. 300 mg, using the MMRM model SAS code as presented above.

For the analysis of time elapsed until the need for rescue medication, a time to event analysis using the Kaplan-Meier survival curve will be performed and the log-rank test will be used to compare the treatment groups. The LIFETEST procedure in SAS will be used to perform this analysis.

#### 4.1 Patient Disposition and Drug Exposure

Patient disposition, based on the Safety population, will be summarized descriptively. Data will include the numbers and percentages of patients who were screened, enrolled, completed the study, and withdrawn (including reasons for withdrawals).

For each patient, the number of doses taken will be computed from the study drug dispensing and accountability eCRFs obtained at each visit. The extent of exposure to study medication, as well as compliance during the study, will be summarized with descriptive statistics.

The number of exposed patients at each study site will be presented by treatment group, and the number of subjects included in each population will be tabulated by treatment group.

#### 4.2 Patient Characteristics

Baseline characteristics will be summarized by mean, standard deviation (SD), median, and minimum and maximum values, for the ITT, PP and the Safety populations. Medical history and prior medications will be summarized descriptively as number of patients and percentage.

### 4.2.1 Demographics

Demographic data (age, sex, ethnicity, and race) will be summarized by treatment group.

### **4.2.2** Medical History

Medical history on current and historical diagnoses and co-morbidities will be coded using the preferred terms (PTs) of the Medical Dictionary for Regulatory Activities (MedDRA), and will be summarized by treatment group.

#### 4.2.3 Prior Medications

Prior medication use will be summarized by treatment group.

#### 4.3 Efficacy Analyses

#### 4.3.1 Primary Efficacy Endpoint

The primary endpoint is the change from baseline to Month 9 in score on the motor examination subscale (Part III) of the MDS-UPDRS. For a detailed definition, see Section 7.1.1 of the study protocol.

The primary efficacy endpoint will be analyzed based on the ITT population. The analysis will be repeated for the PP population as a sensitivity analysis.

The data on the change in Part III score of the MDS-UPDRS from baseline to Month 9 will be summarized by treatment group. The MMRM model will be used to compare the change in score among treatment groups.

#### 4.3.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints are listed below. For detailed definitions, see Section 7.1.2 of the study protocol.

- Change from baseline to Month 9 in total score on the MDS-UPDRS
- Change from baseline to Month 9 in scores on the individual subscales of the MDS-UPDRS: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), and Part IV (motor complications)
- Change from baseline to Month 9 in the combined scores from Parts II and III of the MDS-UPDRS
- Change from baseline to Month 9 in overall cognitive function, as assessed by the Montreal Cognitive Assessment (MoCA) test
- Change from baseline to Month 9 in pharmacodynamics measures of the following oxidative stress biomarkers: total antioxidant status, lipid peroxidation (malondialdehyde), protein carbonyls, 8-OHdG, glutathione, superoxide dismutase
- Change from baseline to Month 9 in pharmacodynamics measures of the following inflammatory factor biomarkers: TNF alpha and IL-6
- Time elapsed until the need for rescue medication

The secondary efficacy endpoints will be analyzed based on the ITT population only.

The data on the changes from baseline to Month 9 in the MDS-UPDRS total score, the Parts I, II, and IV subscale scores, the combined Part II and Part III score, and the MoCA score will be summarized by treatment group. The MMRM model will be used to compare the change in each score between treatment groups.

The data on the changes from baseline to Month 9 in oxidative stress biomarkers and inflammatory factor biomarkers will be summarized by treatment group.

The time elapsed until the need for rescue medication will be presented using the Kaplan-Meier survival curve, and will be compared among the treatment groups using the log-rank test.

#### 4.3.3 Exploratory Efficacy Endpoints

The exploratory objectives of this study are to evaluate whether the potential disease-modifying action of deferiprone is correlated with 1) specific genotypes of enzymes that play a role in Parkinson's disease, and 2) the degree of change from baseline in ceruloplasmin levels and ceruloplasmin ferroxidase activity. The Mechanism of Action (MOA) biomarkers that will be examined are listed below. For detailed definitions, see Section 7.1.3 of the study protocol.

#### The biomarkers are:

- D544E polymorphisms of the glycoprotein ceruloplasmin
- V158M polymorphisms of the enzyme catechol O-methyltransferase (COMT)
- Ceruloplasmin levels (to be analyzed depending on the outcomes of the primary and/or secondary efficacy endpoints)
- Ceruloplasmin ferroxidase activity (to be analyzed depending on the outcomes of the primary and/or secondary efficacy endpoints)

To evaluate the impact of the D544E and V158M genotypes on the treatment effect of deferiprone in Parkinson's disease, subgroup analyses of the data from the two genotypes will be done based on the MMRM analysis performed on the primary endpoint (change from baseline to Month 9 on the Part III score of the MDS-UPDRS), using the ITT population. If there is a treatment effect on the score from other parts of MDS-UPDRS, this analysis will be repeated for those outcomes as well. For details, see Section 4.3.4.

If there is evidence of efficacy based on the primary and/or secondary efficacy endpoints, the data on the change from baseline to Month 9 in ceruloplasmin level and ceruloplasmin ferroxidase activity will be summarized by treatment group. The MMRM model will be used to compare the change in these two biomarkers between treatment groups. Correlation analysis between the change and the primary efficacy endpoint will be performed for each biomarker. These two variables will also be included in the main MMRM model for the primary endpoint, in order to study the relationship between these two MOA biomarkers and the effect of deferiprone.

Correlation analysis of the PD endpoints (change from baseline to Month 9 for biomarkers of interest) and the PK parameters (AUC<sub>0- $\infty$ </sub> and Cmax) will be performed if efficacy is evidenced. This analysis will be performed for the PK/PD population.

#### 4.3.4 Exploratory Analyses/Sensitivity Analysis

If there are unevenly distributed baseline factors among the treatment groups, the effects of those factors on the efficacy measurements will be examined by including them in the MMRM model.

Subgroup analyses will be performed for the ITT population on the following factors: D544E genotype (Aspartate/Aspartate vs. Aspartate/Glutamate) and V158M genotype (Methionine/Methionine vs. Valine/Methionine vs. Valine/Valine). For D544E genotype, Aspartate/Aspartate corresponds to the high metabolizer phenotype (AA) and Aspartate/Glutamate to the low metabolizer phenotype (AT). For the V158M genotypes, the corresponding phenotypes are High COMT Activity, Intermediate COMT Activity, and Low COMT Activity. The analysis results will be presented by the phenotypes for each factor.

Besides analysis for the ITT population, the primary efficacy endpoint will also be analyzed for the PP population as sensitivity analyses.

As a sensitivity analysis, the efficacy data will be re-analyzed with the missing data being imputed as described in section 3.5. The sensitivity analysis will be performed only on the primary efficacy endpoint using the ITT population.

If the blinded review of the efficacy data performed before the breaking of the treatment codes indicates a severe non-normality of the data, an appropriate transformation (for example, log transformation) will be applied to the data, or nonparametric statistical methods based on ranks will be employed, if warranted.

Other exploratory analyses may be performed after examining the planned analyses if they are considered interesting and necessary.

#### 4.4 Safety Analyses

The safety endpoints are listed below. For detailed definitions, see Section 7.2 of the study protocol. Adverse events (AEs)

- Serious adverse events (SAEs)
- Number of discontinuations due to AEs
- Laboratory measures (hematology, blood chemistry, and urinalysis)
- ECG
- Change from baseline in vital signs

- Physical examination
- Assessment of suicidality (as per the Columbia Suicide Severity Rating Scale, C-SSRS)

All safety data collected will be presented in listings and summary tables or graphs to give an overview of the findings. All safety endpoints will be analyzed based on the Safety population.

For laboratory findings, since patients may not attend each study visit within the scheduled time window or may withdraw early, data will be classified into visits according to the time elapsed from the first dose of study medication (date of exposure) to the date of assessment. For biochemistry, the following time windows will be employed:

Month 1 visit: 0 to <1.5 months

Month 2 visit: 1.5 to <2.5 months

Month 3 visit: 2.5 to <3.5 months

Month 4 visit: 3.5 to <4.5 months

Month 5 visit: 4.5 to <5.5 months

Month 6 visit: 5.5 to <7.5 months

Month 9 visit: 7.5 to <10 months

For the weekly hematology visits, data will be classified using half-weeks:

Week 1 visit: 0 to <1.5 weeks

Week 2 visit: 1.5 to <2.5 weeks

. . . .

For other measurements that fall on the same scheduled visits as the efficacy outcomes, such as urinalysis, the rule defined for efficacy outcomes in the beginning of Section 4 will apply.

#### 4.4.1 Adverse Events

A summary table of adverse events by treatment group will include the following information:

- Number of patients exposed to study treatment
- Number of patients experiencing at least one AE
- Number of patients experiencing at least one severe AE
- Number of patients experiencing at least one serious AE
- Number of patients experiencing at least one drug-related AE
- Number of deaths
- Total number of patients withdrawn
- Number of withdrawals due to AEs

Untoward medical occurrences, whether new events or the worsening of severity or frequency of pre-existing conditions, will be coded using MedDRA, and summarized by treatment and by system organ class (SOC) and preferred term (PT). An event will be considered an AE if 1) its start date is on or after the date of the first dose of study medication, 2) the start date is missing and the stop date is on or after the date of the first dose of study medication, or 3) both the start and the stop dates are missing. SAEs that begin within 30 days after the last dose of study medication, and both SAEs and non-serious AEs that are still ongoing for up to 30 days after the last dose, will be included in the database.

Adverse events will be summarized using the total number of events, the total number and percent of patients who experience an AE, and the number and percent of patients who experienced an AE within each SOC (and each PT within an SOC). AEs will also be presented by intensity (mild, moderate, severe), by seriousness (serious, non-serious) and by relationship to study medication (at least possibly related, not related). The number of patients withdrawn and the reasons for withdrawal will also be presented.

To count the number of patients who experienced each AE, a patient who experienced the same AE multiple times will be counted only once for the corresponding preferred term. Similarly, a patient who experienced multiple AEs within the same SOC will be counted only once for that SOC. AEs will be tabulated by presenting the SOCs alphabetically, and within each SOC, the preferred terms will be presented in decreasing order of the total number of patients who experienced each one. In summaries presenting the incidence of AEs by severity, seriousness, and relation to study medication, patients with multiple events coded to a given PT or SOC will be counted only once for that PT or SOC according to the most severe event, the most serious event, or the event with the closest relationship to study medication.

Listing of SAEs and listing of withdrawals due to AEs will be presented. Patient deaths will be listed separately and will be described in narratives.

#### 4.4.2 Vital Signs and Weight

Descriptive statistics (mean, median, standard deviation, minimum and maximum) will be presented at each visit for supine and standing heart rate, supine and standing blood pressure, and weight. Data will also be presented graphically, for examination of possible trends. Change from baseline in these measures (for orthostatic vital signs, the baseline values will be the average of the three sets collected) will be assessed.

#### **4.4.3 12-Lead ECG**

The number and percentage of patients with normal and abnormal ECG results will be provided. Descriptive statistics will be presented for HR, PR, QRS, QT, QTcF, and QTcB.

#### 4.4.4 Biochemistry, Hematology and Urinalysis

Descriptive statistics for each clinical laboratory test will be presented for each scheduled visit. For each test, if multiple measurements are taken on the same visit for a patient, the average value will be used. Using the laboratory's normal ranges, the results will be categorized as low (< lower normal limit), normal (within normal range), or high (> upper normal limit). Shift tables comparing the distributions of these three categories at baseline versus end of treatment will be presented.

Continuous data will also be presented graphically, for examination of possible trends.

Clinically significant abnormalities in laboratory values will be included in the analyses of adverse events.

#### 4.4.5 Concomitant Medications

Medications will be coded using the World Health Organization (WHO) Drug Dictionary. Medications taken during the course of the trial (on or after the first study drug dose and before or on the date of study termination will be considered to be concomitant medications. Medications started after the study termination date will not be reported in tables, but will be presented in patient data listings. Concomitant medications that were used to treat adverse events will be differentiated from others.

Concomitant medications will be summarized according to preferred names only. To count the number of patients who took each type of medication, a patient who took the same medication multiple times will be counted only once for that medication. Medications will be tabulated in decreasing order of the total number of patients who took each one. In addition, the total number of patients to ever take any concomitant medications will be presented.

Concomitant medications will be presented based on the Safety population.

#### 4.4.6 Suicidality

The Columbia Suicide Severity Rating Scale (C-SSRS) is an instrument used to measure suicidal ideation and behavior. For each treatment group, descriptive statistics (frequency and percentage) will be presented for any suicidal ideation and behavior reported by patients at each visit.

### 4.4.7 Treatment Compliance

Compliance will be determined as follows: 1) patients will use the daily diary card to record the number of tablets taken, and 2) at each visit, the investigator or a delegate will inspect the medication containers, whether empty, partly used, or unopened, and will check the number of tablets remaining. Compliance will be calculated by the number of tablets taken divided by the number prescribed, as per the dosing frequency and length of treatment. Compliance at each follow-up visit will be summarized descriptively by treatment group in a table.

#### 5 Listing of Tables and Figures

The summary tables and figures that will be produced based on the statistical analyses detailed in this document are listed bleow. All tables and figures will be presented by treatment group. Tables and figures are numbered following ICH structure, but the final numberings that appear in the clinical study report may be changed if more tables and/or figures are added. The standards used to compile the clinical data will be based on the Study Data Tabulation Model v1.4, SDTM implementation guide v 3.2 as well as controlled terminology v 2017-06-30 from the Clinical Data Interchange Standards Consortium (CDISC). Tables, listings and figures will be programmed using data from the SDTM datasets.

#### Tables Listing:

#### 14.1 Disposition, Demographics and Baseline Data

| Table 14.1.1 | Number of patients in different populations |
|---|---|
| Table 14.1.2 | Subject disposition – Safety population |
| Table 14.1.3 | Subject exposure to study medication – Safety population |
| Table 14.1.4 | Number of patients enrolled by study site – Safety population |
| Table 14.1.5 | Summary of the reasons for not completing the study – Safety |
| | population |
| Table 14.1.6 | Summary of demographics data at baseline – ITT population |
| Table 14.1.6a | Summary of demographics data at baseline – PP population |
| Table 14.1.6b | Summary of demographics data at baseline – Safety population |
| Table 14.1.7 | Summary of baseline characteristics – ITT population |
| Table 14.1.7a | Summary of baseline characteristics – PP population |
| Table 14.1.8 | Medical History – Safety population |
| Table 14.1.9 | Prior Medication – Safety population |

### 14.2 Efficacy Analyses

#### 14.2.1 Primary Efficacy Endpoint

| Table 14.2.1.1 | Change in MDS-UPDRS Part III score at each follow-up visit – ITT |
|---|---|
| | population |
| Table 14.2.1.1a | Change in MDS-UPDRS Part III score at each follow-up visit – PP |
| | population |
| Table 14.2.1.2 | Primary outcome least square mean (LSM) change from baseline to |
| | month 9 from MMRM model – ITT population |
| Table 14.2.1.2a | Primary outcome least square mean (LSM) change from baseline to |
| | month 9 from MMRM model – PP population |
| Table 14.2.1.2s | Primary outcome least square mean (LSM) change from baseline to |
| | month 9 from MMRM model – Sensitivity Analysis population |

| Table 14.2.1.2.1 | Primary outcome least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population and D544E polymorphisms = AA |
|---|---|
| Table 14.2.1.2.2 | 1 7 1 |
| Table 14.2.1.2.3 | Primary outcome least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population and V158M polymorphisms = High COMT Activity |
| Table 14.2.1.2.4 | |
| Table 14.2.1.2.5 | Primary outcome least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population and V158M polymorphisms = Low COMT Activity |
| Table 14.2.1.3 | Dose-response assessment for all efficacy outcomes by linear regression model – ITT population |
| Table 14.2.1.4 | Primary outcome least square mean (LSM) change from baseline to month 9 from MMRM model 2 – ITT population |
| 14.2.2 Secondary Efficacy Endpoints | |
| Table 14.2.2.1 | Change in other MDS-UPDRS scores and MoCA at each follow-up visit – ITT population |
| Table 14.2.2.2 | Change in oxidative stress biomarkers at each follow-up visit – ITT population |
| Table 14.2.2.3 | Change in inflammatory factor biomarkers at each follow-up visit – ITT population |
| Table 14.2.2.4 | Secondary outcomes least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population |
| Table 14.2.2.5 | Secondary outcomes least square mean (LSM) change from baseline to month 9 from MMRM model 2 – ITT population |
| 14.2.3 Exploratory Efficacy Endpoints (only produced if efficacy is evidenced) | |
| Table 14.2.3.1 | Change in MOA biomarkers at each follow-up visit – ITT population |
| Table 14.2.3.2 | MOA biomarkers least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population |
| Table 14.2.3.3 | MOA biomarkers least square mean (LSM) change from baseline to month 9 from MMRM model 2 – ITT population |

## 14.3 Safety Analyses

## 14.3.1 Adverse Events

| Table 14.3.1.1 Table 14.3.1.2 Table 14.3.1.3 Table 14.3.1.4 Table 14.3.1.5 Table 14.3.1.6 | Overall summary of adverse events – safety population Summary of adverse events – safety population All adverse events by severity – safety population All adverse events by seriousness – safety population All adverse events by relatedness to study medication – safety population Summary of most common (>5%) adverse drug reactions – safety population |
|---|---|
| 14.3.2 Hematolo | ogy and Biochemistry and Urinalysis |
| Table 14.3.2.1.1 Table 14.3.2.1.2 Table 14.3.2.2.1 Table 14.3.2.2.2 Table 14.3.2.3.1 | Hematology at each follow-up visit – safety population Shift table comparing three laboratory value categories at baseline and end of study - Hematology – safety population Blood biochemistry at each follow-up visit – safety population Shift table comparing three laboratory value categories at baseline and end of study - Blood biochemistry – safety population Proportions of abnormal urinalysis results in each visit – safety population |
| 14.3.3 Vital Sig | ns and Weight |
| Table 14.3.3.1<br>Table 14.3.3.2<br>Table 14.3.3.3<br>Table 14.3.3.4 | Summary of vital signs at each follow-up visit – safety population Change of vital signs from baseline at each follow-up visit – safety population Summary of weight at each follow-up visit – safety population Change of weight from baseline at each follow-up visit – safety population |
| 14.3.4 12-Lead | ECG |
| Table 14.3.4.1 Table 14.3.4.2 | Summary of 12-lead ECG parameters at each follow-up visit – safety population Proportions of normal and abnormal ECG results in each visit – safety population |
| 14.3.5 Treatment Compliance | |
| Table 14.3.5.1 | Treatment compliance (%) by visit – safety population |
| 14.3.6 Concomitant Medications | |
| Table 14.3.6.1<br>Table 14.3.6.2 | Concomitant Medications – safety population<br>Concomitant PD Medications – safety population |

### 14.3.7 C-SSRS

Table 14.3.7.1 Summary of C-SSRS in each visit – safety population

## Figures Listing:

### 14.2 Efficacy

| Figure 14.2.1.1 | Mean line graph for MDS-UPDRS Part III over visit – ITT population |
|---|---|
| Figure 14.2.1.2 | Mean line graph for MDS-UPDRS Total Score over visit – ITT |
| | population |
| Figure 14.2.1.3 | Mean line graph for MDS-UPDRS Part I over visit – ITT population |
| Figure 14.2.1.4 | Mean line graph for MDS-UPDRS Part II over visit – ITT population |
| Figure 14.2.1.5 | Mean line graph for MDS-UPDRS Part IV over visit – ITT population |
| Figure 14.2.1.6 | Mean line graph for MDS-UPDRS Part II/Part III over visit – ITT |
| | population |
| Figure 14.2.1.7 | Mean line graph for MoCA over visit – ITT population |
| Figure 14.2.1.8 | Mean line graph for Total Antioxidant Status over visit – ITT |
| | population |
| Figure 14.2.1.9 | Mean line graph for Lipid Peroxidation over visit – ITT population |
| Figure 14.2.1.10 | Mean line graph for Protein Carbonyls over visit – ITT population |
| Figure 14.2.1.11 | Mean line graph for 8-OHdG over visit – ITT population |
| Figure 14.2.1.12 | Mean line graph for Glutathione over visit – ITT population |
| Figure 14.2.1.13 | Mean line graph for Superoxide Dismutase over visit – ITT population |
| Figure 14.2.1.14 | Mean line graph for TNF Alpha over visit – ITT population |
| Figure 14.2.1.15 | Mean line graph for IL-6 over visit – ITT population |
| Figure 14.2.2.1 | Kaplan-Meier survival curve for the time to the need for rescue |
| | medication |

## 14.3 Safety

## 14.3.1 Hematology

| Figure 14.3.1.1<br>Figure 14.3.1.2 | Mean line graph for hemoglobin over visit – safety population<br>Mean line graph for total white blood cell (WBC) count over visit – |
|---|---|
| | safety population |
| Figure 14.3.1.3 | Mean line graph for absolute neutrophil count (ANC) over visit – safety population |
| Figure 14.3.1.4 | Mean line graph for platelets over visit – safety population |
| Figure 14.3.1.5 | Mean line graph for mean corpuscular volume (MCV) over visit – safety population |

### 14.3.2 Biochemistry

Figure 14.3.2.1 Mean line graph for serum ferritin over visit – safety population

| Figure 14.3.2.2 | Mean line graph for total protein over visit – safety population |
|---|---|
| Figure 14.3.2.3 | Mean line graph for gamma-glutamyl transferase (GGT) over visit – |
| | safety population |
| Figure 14.3.2.4 | Mean line graph for lactate dehydrogenase (LDH) over visit – safety |
| - | population |
| Figure 14.3.2.5 | Mean line graph for sodium over visit – safety population |
| Figure 14.3.2.6 | Mean line graph for potassium over visit – safety population |
| Figure 14.3.2.7 | Mean line graph for chloride over visit – safety population |
| Figure 14.3.2.8 | Mean line graph for glucose over visit – safety population |
| Figure 14.3.2.9 | Mean line graph for total bilirubin over visit – safety population |
| Figure 14.3.2.10 | Mean line graph for direct bilirubin over visit – safety population |
| Figure 14.3.2.11 | Mean line graph for indirect bilirubin over visit – safety population |
| Figure 14.3.2.12 | Mean line graph for aspartate aminotransferase (AST) over visit – |
| | safety population |
| Figure 14.3.2.13 | Mean line graph for alanine transaminase (ALT) over visit – safety |
| | population |
| Figure 14.3.2.14 | Mean line graph for albumin over visit – safety population |
| Figure 14.3.2.15 | Mean line graph for blood urea nitrogen (BUN) over visit – safety |
| | population |
| Figure 14.3.2.16 | Mean line graph for calcium over visit – safety population |
| Figure 14.3.2.17 | Mean line graph for creatinine over visit – safety population |
| Figure 14.3.2.18 | Mean line graph for uric acid over visit – safety population |
| Figure 14.3.2.19 | Mean line graph for alkaline phosphatase (ALP) over visit – safety |
| | population |
| Figure 14.3.2.20 | Mean line graph for amylase over visit – safety population |
| Figure 14.3.2.21 | Mean line graph for blood iron over visit – safety population |
| Figure 14.3.2.22 | Mean line graph for zinc over visit – safety population |
| Figure 14.3.2.23 | Mean line graph for copper over visit – safety population |
| 14.3.3 Vital Signs | s and Weight |
| Figure 14.3.3.1 | Mean line graph for supine heart rate over visit – safety population |
| | Mean line graph for standing heart rate over visit – safety population |
| Figure 14.3.3.3 | Mean line graph for supine systolic blood pressure over visit – safety |
| C | population |
| Figure 14.3.3.4 | Mean line graph for standing systolic blood pressure over visit – safety |
| $\mathcal{E}$ | population |
| Figure 14.3.3.5 | Mean line graph for supine diastolic blood pressure over visit – safety |
| J | population |
| Figure 14.3.3.6 | Mean line graph for standing diastolic blood pressure over visit – |
| _ | safety population |
| Figure 14.3.3.7 | Mean line graph for weight over visit – safety population |

#### 6 Data Listings

Data listings are numbered following ICH structure. The final numberings for subject data listings in the clinical study report can be changed if more subject data listings are made in the addition to those in the SAP. Collected data have been mapped to SDTM compliant terminology. Randomized subjects who received at least one dose of study drug are included in the listings.

#### Subject Data Listings 16.2

| 16.2.1 Subject Dis | sposition |
|---|---|
| 16.2.1.1<br>16.2.1.2 | Listing of Screening Failures Listing of Disposition |
| 16.2.2 Protocol D | reviations |
| 16.2.2.1 | Listing of Protocol Deviations |
| 16.2.3 Subjects Ex | xcluded from the Efficacy Analysis |
| 16.2.3.1<br>16.2.3.2 | Listing of Randomization Assignment of Subjects to Analysis Sets |
| 16.2.4 Demographic Data and Medical History | |
| 16.2.4.1<br>16.2.4.2<br>16.2.4.3<br>16.2.4.4<br>16.2.4.5 | Listing of Informed Consent Form Listing of Demographics Listing of Parkinson's Disease Diagnosis Listing of Physical Exam Listing of Medical History |
| 16.2.5 Compliance and/or Drug Concentration Data | |
| 16.2.5.1<br>16.2.5.2<br>16.2.5.3 | Listing of Compliance Listing of Exposure Listing of Changes to Exposure |
| 16.2.6 Efficacy D | ata |
| 16.2.6.1 | Listing of Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) scores |
| 16.2.6.2 | Listing of Montreal-Cognitive Assessment (MoCA) |

## 16.2.7 Adverse Events Listing

| 16.2.7.1 | Listing of Medical Events |
|----------|-------------------------------------------|
| 16.2.7.2 | Listing of Adverse Events |
| 16.2.7.3 | Listing of Adverse Drug Reactions |
| 16.2.7.4 | Listing of Serious Adverse Events |
| 16.2.7.5 | Listing of Serious Adverse Drug Reactions |
| 16.2.7.6 | Listing of Withdrawals due to AEs |

## 16.2.8 Listing of Individual Laboratory Measurements by Subjects

| 16.2.8.1 | Listing of Hematology |
|----------|-------------------------------------------|
| 16.2.8.2 | Listing of Biochemistry |
| 16.2.8.3 | Listing of Urinalysis |
| 16.2.8.4 | Listing of Pregnancy Test |
| 16.2.8.5 | Listing of Oxidative Stress Biomarkers |
| 16.2.8.6 | Listing of Inflammatory Factor Biomarkers |

## 16.2.9 Other Listings

| 16.2.9.1 | Listing of Vital Signs |
|-----------|-----------------------------------------------------------------|
| 16.2.9.2 | Listing of Height and Weight |
| 16.2.9.3 | Listing of Concomitant Medications |
| 16.2.9.4 | Listing of Concomitant Medications to treat adverse events |
| 16.2.9.5 | Listing of Medications started after the study termination date |
| 16.2.9.6 | Listing of Columbia Suicide Severity Rating Scale (C-SSRS) |
| 16.2.9.7 | Listing of Telephone Contacts |
| 16.2.9.8 | Listing of Bottle Numbers |
| 16.2.9.9 | Listing of PK Assessment - Informed Consent Form |
| 16.2.9.10 | Listing of PK Assessment |
| 16.2.9.11 | Listing of 12-Lead ECGs |

#### 7 Table Shells

The table shells shown below provide a framework for the display of data in this study. The final tables may not be designed exactly as shown here, but the shells are intended to reflect the general layout of the data that will be included in the clinical study report.

- For descriptive statistics except observation number n, one more decimal place than in the raw data will be presented, and all percentages will be presented with one decimal point unless presented differently in the actual table.
- Note that 'c' in the table shells indicates an alphanumeric character, while 'x' indicates a number from 0 to 9.
- The analysis population is indicated at the end of the table title.
- For tables that are repeated for different populations, those for the PP population will have an 'a' added to the table number, those for the Safety population will have a 'b' added, and those repeated as a sensitivity analysis will have an 's' added: i.e., Table 14.x.x for the ITT population, Table 14.x.xa for the PP population, Table 14.x.xb for the Safety population, and Table 14.x.xs for the sensitivity analysis.

#### Disposition tables

Table 14.1.1 Number of patients in different populations

| Population | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg | Overall |
|------------|---------|--------|--------|--------|---------|---------|
| ITT | XX | xx | XX | xx | XX | XX |
| PP | XX | xx | XX | xx | XX | xx |
| Safety | XX | xx | xx | xx | xx | xx |
| PK/PD | XX | xx | XX | XX | XX | XX |

Table 14.1.2 Subject disposition – Safety population

| | , | Screened= xx | | | | |
|---|---|---|---|---|---|---|
| n (%) | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg | Overall |
| Randomized | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Exposed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawn | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Table 14.1.3 Subject exposure to study medication – Safety population

| | | Group | | | | |
|---|---|---|---|---|---|---|
| | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg | Overall |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Subjects Exposed | xx | XX | xx | xx | xx | xx |
| Total Exposure (person-years) | xxx.x | XXX.X | xxx.x | XXX.X | XXX.X | xxx.x |
| Length of Exposure (years) | | | | | | |
| Mean (SD) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| (Min, Max) | (xx.x,<br>xx.x) | (xx.x,<br>xx.x) | (xx.x,<br>xx.x) | (xx.x,<br>xx.x) | (xx.x,<br>xx.x) | (xx.x,<br>xx.x) |

Table 14.1.4 Number of patients enrolled by study site – Safety population

| Country | Site | | Group | | | | |
|---|---|---|---|---|---|---|---|
| | | Placebo | 300 mg 600 mg 900 mg 1200 mg Overall | | | | |
| Xxx | 000x | XX | XX | XX | XX | XX | XX |
| | | XX | XX | XX | XX | XX | XX |
| Total | X | XX | XX | XX | XX | XX | XX |

Table 14.1.5 Summary of the reasons for not completing the study – Safety population

| | , 21 1110 104 | Group | | | | |
|---|---|---|---|---|---|---|
| | | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) |
| Reason | Detail | n (%) | n (%) | n (%) | n (%) | n (%) |
| A 1 | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Voluntary withdrawal | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Voluntary withdrawar | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow up | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow up | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator desigion | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator decision | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Rescue medication | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| used | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lack of efficacy/<br>worsening of the | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| disease | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Cccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

### Demographics and baseline characteristics tables

Table 14.1.6 Summary of demographics data at baseline – ITT population

| | Group | | | | | | |
|---|---|---|---|---|---|---|---|
| | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) | Overall (N=xx) | <i>p</i> -value <sup>§</sup> |
| Age (years) | | | | | | | 0.xxxx |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| (Minimum, Median, Maximum) | (xx, xx, xx) | (xx, xx, xx) | (xx, xx, xx) | (xx, xx, xx) | (xx, xx, xx) | (xx, xx, xx) | |
| Sex: n (%) | | | | | | | 0.xxxx |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Racial Origin: n (%) | | | | | | | 0.xxxx |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Black | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Native American | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Multi-Racial | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Ethnic Origin: n (%) | | | | | | | 0.xxxx |
| Hispanic/Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

<sup>§</sup> ANOVA for means and Fisher's exact test for percentages

Similar Table 14.1.6a will be based on PP population

Similar Table 14.1.6b will be based on Safety population

Table 14.1.7 Summary of baseline characteristics – ITT population

| | | | | Group | | | |
|---|---|---|---|---|---|---|---|
| | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg | Overall | 1 8 |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | <i>p</i> -value <sup>§</sup> |
| MDS-UPDRS Part III | | | | | | | 0.xxxx |
| n | XX | XX | XX | XX | XX | XX | |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| (Minimum, Maximum) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |
| MDS-UPDRS Total Score | | | | | | | 0.xxxx |
| n | XX | XX | XX | XX | XX | XX | |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| (Minimum, Maximum) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |
| MDS-UPDRS Part I | | | | | | | 0.xxxx |
| n | XX | XX | XX | XX | XX | XX | |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| (Minimum, Maximum) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |
| MDS-UPDRS Part II | | | | | | | 0.xxxx |
| n | XX | XX | XX | XX | XX | XX | |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| (Minimum, Maximum) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |
| MDS-UPDRS Part IV | | | | | | | 0.xxxx |
| n | XX | XX | XX | XX | XX | XX | |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| (Minimum, Maximum) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |

| MDS-UPDRS Part II/Part III | | | | | | | 0.xxxx |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| (Minimum, Maximum) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |
| MoCA | | | | | | | 0.xxxx |
| n | XX | XX | XX | XX | XX | XX | |
| $(Mean \pm SD)$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| (Minimum, Maximum) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |

§ ANOVA

Similar Table 14.1.7a will be based on PP population

Table 14.1.8 Medical History – Safety population

| | Group | | | | | |
|---|---|---|---|---|---|---|
| | Placebo (N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) | Overall (N=xx) |
| Illness/Event by MedDRA Primary System Organ Class and Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ccccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ccccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ccccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ccccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Table 14.1.9 Prior Medication – Safety population

| | Group | | | | | |
|---|---|---|---|---|---|---|
| | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg | Overall |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Drug Name | N Subjects (%) | N Subjects (%) | N Subjects (%) | N Subjects (%) | N Subjects (%) | N Subjects (%) |
| Preferred Name | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ccccc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
## Efficacy outcomes tables

Table 14.2.1.1 Change in MDS-UPDRS Part III score at each follow-up visit – ITT population

| | Visit | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) |
|---|---|---|---|---|---|---|
| | Baseline | xx | XX | XX | XX | XX |
| | | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| MDS-UPDRS | Month 3 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Part III score | | XX.X | XX.X | XX.X | XX.X | XX.X |
| n | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Mean (SD) | Change at | XX | XX | XX | XX | XX |
| Median | Month 6 | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| (Min, Max) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| | Month 9 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |

Similar Table 14.2.1.1a will be based on PP population

Table 14.2.1.2 Primary outcome least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population

| Outcome | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 300 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 600 mg<br>(N=xx) | 600 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 900 mg<br>(N=xx) | 900 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 1200 mg<br>(N=xx) | 1200 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value |
|---|---|---|---|---|---|---|---|---|---|
| MDS-<br>UPDRS<br>Part III<br>score<br>LSM<br>(SE) | xx.x<br>(xx.x) | xx.x<br>(xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | xx.x<br>(xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | xx.x<br>(xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | xx.x<br>(xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx |

Similar Table 14.2.1.2a will be based on PP population

Similar Table 14.2.1.2s will be based on sensitivity analysis population (ITT with missing data imputation)

Similar Tables 14.2.1.2.1 and 14.2.1.2.2 will be based on ITT population and D544E polymorphisms (AA vs. AT) Similar Tables 14.2.1.2.3, 14.2.1.2.4 and 14.2.1.2.5 will be based on ITT population and V158M polymorphisms (High vs. Intermediate vs. Low COMT Activity)

Table 14.2.1.3 Dose-response assessment for all efficacy outcomes by linear regression model – ITT population

| Dependent variable | Regression Slope | P - value |
|---|---|---|
| MDS-UPDRS Part III score | X.XX | 0.xxxxx |
| Repeat for other secondary and exploratory efficacy endpoints | | |

Table 14.2.1.4 Primary outcome least square mean (LSM) change from baseline to month 9 from MMRM model 2 – ITT

population

| Outcome | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 600 mg –<br>300 mg<br>LSM<br>(95% CI)<br>p-value | 900 mg<br>(N=xx) | 900 mg –<br>600 mg<br>LSM<br>(95% CI)<br>p-value | 1200 mg<br>(N=xx) | 1200 mg –<br>900 mg<br>LSM<br>(95% CI)<br>p-value |
|---|---|---|---|---|---|---|---|---|
| MDS-<br>UPDRS Part<br>III score<br>LSM<br>(SE) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx | xx.x (xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx | xx.x (xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx |

Note: only produced when there is a significant dose-response relationship in treatment effect

Table 14.2.2.1 Change in other MDS-UPDRS scores and MoCA at each follow-up visit – ITT population

| 14.2.2.1 C | nange in omer | | ores and MoCA at | | | |
|---|---|---|---|---|---|---|
| | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
| | VISIC | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| MDS-UPDRS | Month 3 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Total score | | XX.X | XX.X | XX.X | XX.X | XX.X |
| n | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Mean (SD) | Change at | XX | XX | XX | XX | XX |
| Median | Month 6 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| (Min, Max) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| | Month 9 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for<br>MDS-UPDRS | | | | | | |
| Part I, II, IV | | | | | | |
| and sum of Part | | | | | | |
| II/III score and | | | | | | |
| MoCA | | | | | | |

Table 14.2.2.2 Change in oxidative stress biomarkers at each follow-up visit – ITT population

| Table 14.2.2.2 C | nange in oxida | ative stress bioma | rkers at each follo | w-up visit – 11 1 | _ • | _ |
|---|---|---|---|---|---|---|
| | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
| | VISIT | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Total | Change at | XX | XX | XX | XX | XX |
| Antioxidant | Month 3 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Status | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| n | Change at | XX | XX | XX | XX | XX |
| Mean (SD) | Month 6 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| (Min, Max) | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| | Month 9 | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for | | | | | | |
| Lipid | | | | | | |
| Peroxidation, | | | | | | |
| Protein | | | | | | |
| Carbonyls, 8- | | | | | | |
| OHdG, | | | | | | |
| Glutathione, | | | | | | |
| and Superoxide | | | | | | |
| Dismutase | | | | | | |

Table 14.2.2.3 Change in inflammatory factor biomarkers at each follow-up visit – ITT population

| | | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|---|
| | Visit | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| TNF Alpha | Month 3 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| n | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Mean (SD) | Change at | XX | XX | XX | XX | XX |
| Median | Month 6 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| (Min, Max) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| | Month 9 | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for IL-6 | | | | | | |

Table 14.2.2.4 Secondary outcomes least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population

| population | | | T | 1 | 1 | 1 | | 1 | 1 |
|---|---|---|---|---|---|---|---|---|---|
| Outcome | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 300 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 600 mg<br>(N=xx) | 600 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 900 mg<br>(N=xx) | 900 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 1200 mg<br>(N=xx) | 1200 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value |
| MDS-<br>UPDRS<br>Total<br>score<br>LSM<br>(SE) | XX.X<br>(XX.X) | xx.x<br>(xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | XX.X<br>(XX.X) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | XX.X<br>(XX.X) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | XX.X<br>(XX.X) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx |
| Repeat for<br>MDS-<br>UPDRS<br>Part I, II,<br>IV and<br>sum of<br>Part II/III<br>score and<br>MoCA | | | | | | | | | |

Table 14.2.2.5 Secondary outcomes least square mean (LSM) change from baseline to month 9 from MMRM model 2 – ITT

population

| population | 1 | 1 | T | T | 1 | 1 | 1 | , , |
|---|---|---|---|---|---|---|---|---|
| Outcome | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 600 mg –<br>300 mg<br>LSM<br>(95% CI)<br>p-value | 900 mg<br>(N=xx) | 900 mg –<br>600 mg<br>LSM<br>(95% CI)<br>p-value | 1200 mg<br>(N=xx) | 1200 mg –<br>900 mg<br>LSM<br>(95% CI)<br>p-value |
| MDS-<br>UPDRS<br>Total score<br>LSM<br>(SE) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx | xx.x (xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx | xx.x (xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx |
| Repeat for<br>MDS-<br>UPDRS<br>Part I, II, IV<br>and sum of<br>Part II/III<br>score and<br>MoCA | | | | | | | | |

Note: only produced when there is a significant dose-response relationship in treatment effect

Table 14.2.3.1 Change in MOA biomarkers at each follow-up visit – ITT population

| | | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|---|
| | Visit | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| Ceruloplasmin | Month 3 | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| n | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Mean (SD) | Change at | XX | XX | XX | XX | XX |
| Median | Month 6 | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) |
| (Min, Max) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Change at | XX | XX | XX | XX | XX |
| | Month 9 | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for | | | ••• | | ••• | |
| Ceruloplasmin | | | | | | |
| ferroxidase | | | | | | |
| activity | | | | | | |

Note: only produced if efficacy is evidenced

Table 14.2.3.2 MOA biomarkers least square mean (LSM) change from baseline to month 9 from MMRM model – ITT population

| Outcome | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 300 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 600 mg<br>(N=xx) | 600 mg - Placebo LSM (95% CI) p-value | 900 mg<br>(N=xx) | 900 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value | 1200 mg<br>(N=xx) | 1200 mg -<br>Placebo<br>LSM<br>(95% CI)<br>p-value |
|---|---|---|---|---|---|---|---|---|---|
| Ceruloplasmin<br>LSM<br>(SE) | xx.x<br>(xx.x) | xx.x<br>(xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | XX.X<br>(XX.X) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | xx.x<br>(xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | xx.x<br>(xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx |
| Repeat for<br>Ceruloplasmin<br>ferroxidase<br>activity | | | | | | | | | |

Note: only produced if efficacy is evidenced

Table 14.2.3.3 MOA biomarkers least square mean (LSM) change from baseline to month 9 from MMRM model 2 – ITT population

| Outcome | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 600 mg –<br>300 mg<br>LSM<br>(95% CI)<br>p-value | 900 mg<br>(N=xx) | 900 mg –<br>600 mg<br>LSM<br>(95% CI)<br>p-value | 1200 mg<br>(N=xx) | 1200 mg –<br>900 mg<br>LSM<br>(95% CI)<br>p-value |
|---|---|---|---|---|---|---|---|---|
| Ceruloplasmin<br>LSM<br>(SE) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | xx.x (xx.x) | xx.x<br>(xx.x,<br>xx.x)<br>0.xxxx | xx.x (xx.x) | xx.x<br>(xx.x, xx.x)<br>0.xxxx |
| Repeat for<br>Ceruloplasmin<br>ferroxidase<br>activity | | | | | | | | |

Note: only produced if efficacy is evidenced and when there is a significant dose-response relationship in treatment effect

## Safety outcomes tables

Table 14.3.1.1 Overall summary of adverse events – safety population

| | | Т | reatment Gro | oup | |
|---|---|---|---|---|---|
| | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Number of subjects with at least one AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of subjects with at least one SAE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of subjects with at least one severe AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of subjects with at least one ADR | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of deaths | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of subject withdrawn | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of subject withdrawals due to AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Table 14.3.1.2 Summary of adverse events – safety population

| | Placebo | | 300 mg | | Repeat for 600 mg, 900 mg, and 1200 mg | |
|---|---|---|---|---|---|---|
| | Exposure (subje | ct-years): x.xx | Exposure (subject | z-years): x.xx | Exposure (subject | t-years): x.xx |
| | Total Subjects E | Total Subjects Exposed: xx | | posed: xx | Total Subjects Ex | posed: xx |
| | Total Events: xx | Total Events: xxx | | | Total Events: xxx | |
| | Total Subjects R | eporting: xx (xx%) | Total Subjects Reporting: xx (xx%) | | Total Subjects Reporting: xx (xx | |
| System Organ Class Preferred Term | N Subjects (%) | N Events<br>(Rate/100 patient<br>years) | N Subjects (%) | N Events<br>(Rate/100 patient<br>years) | N Subjects (%) | N Events<br>(Rate/100 patient<br>years) |
| CCCCCC | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) |
| Ccccc | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) |
| Ccccc | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) |
| Ccccc | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) |
| | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) | x (x.x) | x (x.xx) |

Table 14.3.1.3 All adverse events by severity – safety population

| | Placebo $(N = xx)$ | | | | 300 mg $(N = xx)$ | | | Repeat for 600 mg, 900 mg, and 1200 mg | |
|---|---|---|---|---|---|---|---|---|---|
| | Mild | Moderate | Mild | Moderate | Severe | Severe | Mild | Moderate | Severe |
| Any Adverse Event | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| System Organ Class 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Preferred Term 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Continue for all SOC and PTs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| SOCs and Preferred<br>terms sorted<br>alphabetically | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Table 14.3.1.4 All adverse events by seriousness – safety population

| | Placebo $(N = xx)$ | | | mg = xx) | Repeat for 600 mg, 900 mg,<br>and 1200 mg | |
|---|---|---|---|---|---|---|
| | Non-serious | Serious | Non-serious | Serious | Non-serious | Serious |
| Any Adverse Event | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| System Organ Class 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Preferred Term 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Continue for all SOC and PTs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| SOCs and Preferred terms sorted alphabetically | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Table 14.3.1.5 All adverse events by relatedness to study medication – safety population

| | Placebo (N = xx) | | | ) mg<br>= xx) | Repeat for 600 mg, 900 mg,<br>and 1200 mg<br>(N = xx) | |
|---|---|---|---|---|---|---|
| | Related | Unrelated | Related | Unrelated | Related | Unrelated |
| Any Adverse Event | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| System Organ Class 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Preferred Term 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Continue for all SOC and | | | | | | |
| Continue for all SOC and<br>PTs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| SOCs and Preferred terms sorted alphabetically | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Table 14.3.1.6 Summary of most common (>5%) adverse drug reactions – safety population

| | | Placebo | | | 300 mg | | Repeat for | r 600 mg, 900 mg, | and 1200 mg |
|---|---|---|---|---|---|---|---|---|---|
| | | (N = xx) | | | (N = xx) | | | (N = xx) | |
| | n (%) | Time to onset<br>(Days)<br>Mean (SD)<br>Median<br>(Min, Max) | Duration<br>(Days)<br>Mean (SD)<br>Median<br>(Min, Max) | n (%) | Time to onset<br>(Days)<br>Mean (SD)<br>Median<br>(Min, Max) | Duration<br>(Days)<br>Mean (SD)<br>Median<br>(Min, Max) | n (%) | Time to onset<br>(Days)<br>Mean (SD)<br>Median<br>(Min, Max) | Duration<br>(Days)<br>Mean (SD)<br>Median<br>(Min, Max) |
| Any Adverse Event | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) |
| System Organ Class 1 | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) |
| Preferred Term 1 | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) |
| Continue for all SOC and PTs | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) |
| SOCs and Preferred terms<br>sorted alphabetically | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>(xx%) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx.xx (xx.x)<br>xx.x<br>(xx.x, xx.x) |

Table 14.3.2.1.1 Hematology at each follow-up visit – safety population

| 14616 1 1.5.2.1.1 1161114661 | T at each fello | w-up visit – saicty | | 600 | 000 | 1200 |
|---|---|---|---|---|---|---|
| Test | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
| Test | VISIT | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Month 1 | XX | XX | XX | XX | XX |
| Hemoglobin (g/L) | | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| n | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean (SD) | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Median (SD) | Month 2 | XX | XX | XX | XX | XX |
| (Min, Max) | | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| (wiiii, wax) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Repeat for | | | | | |
| | Month 3, 4, 5, | | | | | |
| | 6 and 9 visits | | | | | |
| Repeat for other | | | | | | |
| hematology parameters | | | | | | |

Table 14.3.2.1.2 Shift table comparing three laboratory value categories at baseline and end of study: Hematology – safety population

| I -1 T | T | Danatina | | End of stud | ly | T-4-1 |
|---|---|---|---|---|---|---|
| Laboratory Test | Treatment | Baseline | Low | Normal | High | Total |
| | | Low | XX | XX | XX | XX |
| | Placebo | Normal | XX | XX | XX | XX |
| | Placedo | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | | Low | XX | XX | XX | XX |
| | 300 mg | Normal | XX | XX | XX | XX |
| | 300 mg | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | 600 mg | Low | XX | XX | XX | XX |
| Hemoglobin | | Normal | XX | XX | XX | XX |
| | | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | 000 | Low | XX | XX | XX | XX |
| | | Normal | XX | XX | XX | XX |
| | 900 mg | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | | Low | XX | XX | XX | XX |
| | 1200 ma | Normal | XX | XX | XX | XX |
| | 1200 mg | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| Repeat for other tests of interest | | | | | | |

Table 14.3.2.2.1 Blood biochemistry at each follow-up visit – safety population

| 1 autc 14.3.2.2.1 Blood blo | | 1 | | | 000 | 1200 |
|---|---|---|---|---|---|---|
| Test | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
| 1051 | V 151t | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Month 1 | XX | XX | XX | XX | XX |
| Zinc (g/L) | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) |
| n | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean (SD) | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Median | Month 2 | XX | XX | XX | XX | XX |
| (Min, Max) | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) |
| (Willi, Widx) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Repeat for | | | | | |
| | Month 3, 4, 5, | | | | | |
| | 6 and 9 visits | | | | | |
| Repeat for other | | | | | | |
| biochemistry parameters | | | | | | |

Table 14.3.2.2.2 Shift table comparing three laboratory value categories at baseline and end of study: Blood biochemistry – safety population

| Laboratory Tost | Trantmant | Dagalina | | End of stud | ly | Total |
|---|---|---|---|---|---|---|
| Laboratory Test | Treatment | Baseline | Low | Normal | High | Total |
| | | Low | XX | XX | XX | XX |
| | Placebo | Normal | XX | XX | XX | XX |
| | Flacebo | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | | Low | XX | XX | XX | XX |
| | 200 m a | Normal | XX | XX | XX | XX |
| | 300 mg | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | 600 mg | Low | XX | XX | XX | XX |
| Zinc | | Normal | XX | XX | XX | XX |
| | | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | | Low | XX | XX | XX | XX |
| | 000 | Normal | XX | XX | XX | XX |
| | 900 mg | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| | | Low | XX | XX | XX | XX |
| | 1200 mg | Normal | XX | XX | XX | XX |
| 12 | 1200 mg | High | XX | XX | XX | XX |
| | | Total | XX | XX | XX | XX |
| Repeat for other tests of interest | | | | | | |

Table 14.3.2.3.1 Proportions of abnormal urinalysis results in each visit – safety population

| Test | Visit | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) |
|---|---|---|---|---|---|---|
| A1 111: 1 : | Baseline | xx<br>xx (xx.x) | xx<br>xx (xx.x) | xx<br>xx (xx.x) | xx<br>xx (xx.x) | xx<br>xx (xx.x) |
| Abnormal Urinalysis<br>n<br>Abnormal (n (%)) | Month 3 | xx<br>xx (xx.x) | xx<br>xx (xx.x) | xx<br>xx (xx.x) | xx<br>xx (xx.x) | xx<br>xx (xx.x) |
| | Repeat for Month 6 and 9 visits | | | | | |

Table 14.3.3.1 Summary of vital signs at each follow-up visit – safety population

| Test | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|---|
| 1000 | V 1510 | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Month 1 | XX | XX | XX | XX | XX |
| Supine Heart Rate | | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| n | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean (SD) | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Median | Month 2 | XX | XX | XX | XX | XX |
| (Min, Max) | | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| (Willi, Wax) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Repeat for | | | | | |
| | Month 3, 4, 5, | | | | | |
| | 6 and 9 visits | | | | | |
| Repeat for standing | | | | | | |
| heart rate, supine and | | | | | | |
| standing blood pressure | | | | | | |

Table 14.3.3.2 Change of vital signs from baseline at each follow-up visit – safety population

| Table 14.3.3.2 Change of vital signs from basefine at each follow-up visit – safety population | | | | | | |
|---|---|---|---|---|---|---|
| Test | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
| 1031 | V 151t | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Month 1 | XX | XX | XX | XX | XX |
| Change in Supine Heart | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Rate | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| n<br>Mean (SD) | | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| Median (SD) | Month 2 | XX | XX | XX | XX | XX |
| (Min, Max) | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| <i>p</i> -value | | XX.X | XX.X | XX.X | XX.X | XX.X |
| p-value | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |
| | Repeat for | | | | | |
| | Month 3, 4, 5, | | | | | |
| | 6 and 9 visits | | | | | |
| Repeat for standing | | | | | | |
| heart rate, supine and | | | | | | |
| standing blood pressure | | | | | | |

Table 14.3.3.3 Summary of weight at each follow-up visit – safety population

| Test | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|---|
| Test | VISIL | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Weight | | XX.X | XX.X | XX.X | XX.X | XX.X |
| n | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Mean (SD) | Month 9 | XX | XX | XX | XX | XX |
| Median | | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| (Min, Max) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |

Table 14.3.3.4 Change of weight from baseline at each follow-up visit – safety population

| Test | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|---|
| Test | VISIT | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Change in weight | | XX.X | XX.X | XX.X | XX.X | XX.X |
| n | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Mean (SD) | Month 9 | XX | XX | XX | XX | XX |
| Median | | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| (Min, Max) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| <i>p</i> -value | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx | 0.xxxx |

Table 14.3.4.1 Summary of 12-lead ECG parameters at each follow-up visit – safety population

| Test | Visit | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) |
|---|---|---|---|---|---|---|
| Heart Rate (bpm) n Mean (SD) Median (Min, Max) | Baseline Month 9 | xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x)<br>xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x)<br>xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x)<br>xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x)<br>xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x) | xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x)<br>xx<br>xx.x (xx.x)<br>xx.x<br>(xx.x, xx.x) |
| Repeat for PR Interval,<br>QRS Interval, QT<br>Interval, QTcB<br>Interval, and QTcF<br>Interval | | | | | | |

Table 14.3.4.2 Proportions of normal and abnormal ECG results in each visit – safety population

| Test | Visit | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) |
|---|---|---|---|---|---|---|
| ECG | Baseline | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) |
| n<br>Abnormal (n (%))<br>Normal (n (%)) | Month 9 | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) | XX<br>XX (XX.X)<br>XX (XX.X) | xx<br>xx (xx.x)<br>xx (xx.x) | XX<br>XX (XX.X)<br>XX (XX.X) |

Table 14.3.5.1 Treatment compliance (%) by visit – safety population

| Test | Visit | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|---|
| Test | VISIT | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | Baseline | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Month 1 | XX | XX | XX | XX | XX |
| Compliance (%) | | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| 1 , | | XX.X | XX.X | XX.X | XX.X | XX.X |
| n<br>Mean (SD)<br>Median<br>(Min, Max) | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Month 2 | XX | XX | XX | XX | XX |
| | | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Repeat for | | | | | |
| | Month 3, 4, 5, | | | | | |
| | 6 and 9 visits | | | | | |

Table 14.3.6.1 Concomitant Medications – safety population

| | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|
| | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx |
| | Total Subjects Exposed: xx | Total Subjects Exposed: xx | Total Subjects Exposed: xx | Total Subjects Exposed: xx | Total Subjects Exposed: xx |
| | Total Subjects Reporting: xx | Total Subjects Reporting: xx | Total Subjects Reporting: xx | Total Subjects Reporting: xx | Total Subjects Reporting: xx |
| Drug Name | | | | | |
| Preferred Name | N Subjects (%) | N Subjects (%) | N Subjects (%) | N Subjects (%) | N Subjects (%) |
| Ccccc | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Ccccc | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Table 14.3.6.2 Concomitant PD Medications – safety population

| | Placebo | 300 mg | 600 mg | 900 mg | 1200 mg |
|---|---|---|---|---|---|
| | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx | Exposure (subject-years): x.xx |
| | Total Subjects Exposed: xx | Total Subjects Exposed: xx | Total Subjects Exposed: xx | Total Subjects Exposed: xx | Total Subjects Exposed: xx |
| | Total Subjects Reporting: xx | Total Subjects Reporting: xx | Total Subjects Reporting: xx | Total Subjects Reporting: xx | Total Subjects Reporting: xx |
| Drug Name | | | | | |
| Preferred Name | N Subjects (%) | N Subjects (%) | N Subjects (%) | N Subjects (%) | N Subjects (%) |
| Ccccc | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Ccccc | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Table 14.3.7.1 Summary of C-SSRS in each visit – safety population

| Test | Visit | Placebo<br>(N=xx) | 300 mg<br>(N=xx) | 600 mg<br>(N=xx) | 900 mg<br>(N=xx) | 1200 mg<br>(N=xx) |
|---|---|---|---|---|---|---|
| | Baseline | XX | XX | XX | XX | XX |
| | (Lifetime) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| | Baseline (past | XX | XX | XX | XX | XX |
| C-SSRS | 9 months) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| n | Month 1 | XX | XX | XX | XX | XX |
| Any Suicidal Ideation (n (%)) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Suicidal Behavior (n (%)) | Repeat for | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Month 2, 3, 4, | ••• | ••• | ••• | ••• | |
| | 5, 6 and 9 | | | | | |
| | visits | | | | | |